CLINICAL TRIAL: NCT02965976
Title: Double-Arm, Randomized Study of Botulinum Toxin Injection as a Pyloric Drainage Procedure for Minimally Invasive Esophagectomy (Phase II)
Brief Title: Botulinum Toxin Type A in Preventing Complications After Surgery in Patients With Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: I 283516; NCI-2016-01568 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 283516 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-01

CONDITIONS: Esophageal Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA; incobotulinumtoxinA; Esophagectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (botulinum toxin type A, esophagectomy) (Experimental): Patients receive botulinum toxin type A injection IM while undergoing standard minimally invasive esophagectomy.
  Interventions: Biological: Botulinum Toxin Type A; Procedure: Esophagectomy; Other: Quality-of-Life Assessment
- Arm II (esophagectomy) (Active Comparator): Patients undergo standard minimally invasive esophagectomy.
  Interventions: Procedure: Esophagectomy; Other: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Botulinum Toxin Type A — Given IM
  Other Names: AbobotulinumtoxinA; Botox; Botox Cosmetic; Botulinum A Toxin; Botulinum Neurotoxin Type A; Botulinum Toxin A; BTX-A; Dysport; EvabotulinumtoxinA; IncobotulinumtoxinA; OnabotulinumtoxinA; Onaclostox; Xeomin
  Arms: Arm I (botulinum toxin type A, esophagectomy)
Procedure: Esophagectomy — Undergo esophagectomy
  Other Names: excision of the esophagus
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase II trial studies how well botulinum toxin type A works in preventing complication after surgery in patients with esophageal cancer. Botulinum toxin type A may cause less complications of nausea and vomiting after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if intra-pyloric botulinum toxin type A (botulinum toxin) injection (Botox) during a minimally invasive esophagectomy decreases postoperative occurrence of delayed gastric emptying.

SECONDARY OBJECTIVES:

I. Determine if intra-pyloric botulinum toxin injection during a minimally invasive esophagectomy reduces the number of repeat procedures for delayed gastric emptying within 90 days.

II. Determine if intra-pyloric botulinum toxin injection during a minimally invasive esophagectomy decreases time to oral intake meeting 100% of nutritional requirements.

III. Determine if intra-pyloric botulinum toxin injection during a minimally invasive esophagectomy reduces the incidence of pulmonary complications directly related to delayed gastric emptying.

IV. Determine if intra-pyloric botulinum toxin injection during a minimally invasive esophagectomy reduces hospital length of stay related to delayed gastric emptying.

V. Determine if intra-pyloric botulinum toxin injection during a minimally invasive esophagectomy increases patient quality of life.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive botulinum toxin type A injection intramuscularly (IM) while undergoing standard minimally invasive esophagectomy.

ARM II: Patients undergo standard minimally invasive esophagectomy.

After completion of study treatment, patients are followed up at 2, 3-4, and 6-8 weeks, and at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Esophageal carcinoma, undergoing minimally invasive esophagectomy with intrathoracic anastomosis
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients who have a history of gastrointestinal dysmotility or functional gastroparesis, including diabetic gastroparesis, central and peripheral nervous system disorders, renal failure, medication side effects, including chronic dependence of promotility agents, anticholinergic antispasmodic agents, or chronic narcotic use over 2 years due to non-cancer causes
* Patients who have a history of previous gastric or duodenal surgery
* Patients who have a history of duodenal ulcer or duodenal fibrosis
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Allergy to botulinum toxin and/or egg
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moshim Kukar, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Botulinum Toxin Type A, Esophagectomy) | Arm II (Esophagectomy)
Started | 15 | 17
Completed | 13 | 17
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Botulinum Toxin Type A, Esophagectomy) | Arm II (Esophagectomy) | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (8.0) | 61.2 (11.0) | 62.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 15 | 15 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 16 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 32
Neoadjuvant Chemotherapy Status [Count of Participants; unit: Participants]
  Yes | 14 | 16 | 30
  No | 1 | 1 | 2
Self Reported Smoking Status [Count of Participants; unit: Participants]
  Never Smoked | 0 | 0 | 0
  Former Smoker | 15 | 16 | 31
  Current Smoker | 0 | 1 | 1
Diabetes Status [Count of Participants; unit: Participants]
  Yes | 4 | 5 | 9
  No | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Delayed Gastric Emptying Assessed Radiographically by Nuclear Medicine Emptying Study
Description: Will be assessed using the intent-to-treat principle and a one-sided Cochran-Mantel-Haenszel (CMH) test.
Time Frame: Up to day 21
Population: In Arm I, 2 patients withdrew prior to assessment of primary and secondary outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Botulinum Toxin Type A, Esophagectomy) | Arm II (Esophagectomy)
Number analyzed (Participants) | 13 | 17
Participants
  Delayed Gastric Emptying | 12 | 14
  No Delayed Gastric Emptying | 1 | 3
Statistical Analysis 1: Comparison: Arm I (Botulinum Toxin Type A, Esophagectomy) vs Arm II (Esophagectomy); Test type: Superiority; p = 0.773, Cochran-Mantel-Haenszel

2. Secondary Outcome: Delayed Gastric Emptying Assessed Radiographically by Gastrografin Swallow OR CT Esophagram
Description: Delayed gastric emptying assessed Radiographically by Gastrografin Swallow OR CT Esophagram at day 7. Will be compared between treatment arms using the two-sided CMH exact test.
Time Frame: At day 7
Population: 2 patients in Arm I withdrew prior to any assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Botulinum Toxin Type A, Esophagectomy) | Arm II (Esophagectomy)
Number analyzed (Participants) | 13 | 17
Participants
  Delayed gastric Emptying | 12 | 14
  No Delayed Gastric Emptying | 1 | 3
Statistical Analysis 1: Comparison: Arm I (Botulinum Toxin Type A, Esophagectomy) vs Arm II (Esophagectomy); Test type: Superiority; p = 0.773, Cochran-Mantel-Haenszel

3. Secondary Outcome: Gastrointestinal and Nutritional Status Including Days to Resumption of Oral Feeding as Assessed by Dietician
Description: The days to resumption of oral feeding are calculated based on return to a solid diet. Will be compared between treatment arms using the two sided independent-sample, stratified T-test.
Time Frame: Up to day 35
Population: 2 patients in Arm I withdrew prior to study assessments. Data were not captured and is unavailable for 1 patient in Arm I and 4 patients in Arm II.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm I (Botulinum Toxin Type A, Esophagectomy) | Arm II (Esophagectomy)
Number analyzed (Participants) | 10 | 13
days | 22.6 (4.7) | 27 (16.2)
Statistical Analysis 1: Comparison: Arm I (Botulinum Toxin Type A, Esophagectomy) vs Arm II (Esophagectomy); Test type: Superiority; p = 0.368, t-test, 2 sided

4. Secondary Outcome: Hospital Length of Stay Attributed to Delayed Gastric Emptying
Description: The total length of stay is calculated as the difference between the date of procedure and date of discharge. Will be compared between treatment arms using the two sided independent-sample, stratified T-test.
Time Frame: Up to 90 days
Population: 2 participants in arm I withdrew prior to any study assessments. Data were not captured and unavailable for 1 patient in Arm I and 1 patient in Arm II.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm I (Botulinum Toxin Type A, Esophagectomy) | Arm II (Esophagectomy)
Number analyzed (Participants) | 10 | 16
days | 7.9 (4.2) | 8.1 (1.9)
Statistical Analysis 1: Comparison: Arm I (Botulinum Toxin Type A, Esophagectomy) vs Arm II (Esophagectomy); Test type: Superiority; p = 0.987, t-test, 2 sided

5. Secondary Outcome: Secondary Procedure Due to Delayed Gastric Emptying
Description: The rate of secondary procedures (within 90 days) will be compared between treatment arms using a one-sided CMH exact test.
Time Frame: Up to 90 days
Population: 2 participants in arm I withdrew prior to any study assessments. Data were not captured and unavailable for 2 patients in Arm I and 2 patients in Arm II.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Botulinum Toxin Type A, Esophagectomy) | Arm II (Esophagectomy)
Number analyzed (Participants) | 11 | 15
Participants
  Reoperation | 1 | 0
  No Reoperation | 10 | 15
Statistical Analysis 1: Comparison: Arm I (Botulinum Toxin Type A, Esophagectomy) vs Arm II (Esophagectomy); Test type: Superiority; p = 0.423, Cochran-Mantel-Haenszel

6. Secondary Outcome: Pulmonary Events Directly Related to Delayed Gastric Emptying as Assessed by Operating Surgeon
Description: The rate of post-operative pulmonary events will be compared between treatment arms using the two-sided CMH exact test.
Time Frame: Up to day 90
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Botulinum Toxin Type A, Esophagectomy) | Arm II (Esophagectomy)
Number analyzed (Participants) | 12 | 16
Participants
  Pulmonary Complication | 3 | 3
  No Pulmonary Complication | 9 | 13
Statistical Analysis 1: Comparison: Arm I (Botulinum Toxin Type A, Esophagectomy) vs Arm II (Esophagectomy); Test type: Superiority; p = 1.000, Cochran-Mantel-Haenszel

7. Secondary Outcome: Quality of Life Score as Assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 OES18
Description: Will be compared between treatment arms using the two sided independent-sample, stratified T-test.
Time Frame: Up to day 90
Population: The quality of life data were not captured.
Arm/Group | Arm I (Botulinum Toxin Type A, Esophagectomy) | Arm II (Esophagectomy)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 90 days after surgery.
Arm/Group | Arm I (Botulinum Toxin Type A, Esophagectomy) | Arm II (Esophagectomy)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/15 | 2/17
Other Adverse Events (participants affected / at risk) | 8/15 | 10/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Botulinum Toxin Type A, Esophagectomy) (N=15) | Arm II (Esophagectomy) (N=17)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Postoperative thoracic procedure complication (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Botulinum Toxin Type A, Esophagectomy) (N=15) | Arm II (Esophagectomy) (N=17)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chest pain (Cardiac disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (8)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 5 (5)
Fatigue (General disorders) | 3 (4) | 4 (4)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4)
Weakness (General disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT02965976/Prot_SAP_000.pdf